CLINICAL TRIAL: NCT04137653
Title: Treatment of Triple-negative Breast Cancer With Albumin-bound Paclitaxel as Neoadjuvant Therapy: a Prospective Randomized Controlled Clinical Trial
Brief Title: Treatment of Triple-negative Breast Cancer With Albumin-bound Paclitaxel as Neoadjuvant Therapy: a Prospective RCT
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Shengjing Hospital (Other)
Responsible Party: Principal Investigator, Caigang Liu, Principal Investigator, Shengjing Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Shengjing-LCG004
Record Dates: First submitted 2019-10-22; First posted 2019-10-24 (Actual); Last update posted 2021-07-20 (Actual); Status verified 2021-07

CONDITIONS: Breast Cancer
Keywords: paclitaxel; albumin-bound paclitaxel; neoadjuvant therapy
MeSH Terms: conditions — Breast Neoplasms | interventions — CP protocol

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- nab-Paclitaxel group (Experimental): 749 patients will be assigned into nab-Paclitaxel group.
  Interventions: Drug: nab-Paclitaxel+carboplatin
- paclitaxel group (Active Comparator): 749 patients will be assigned into paclitaxel group
  Interventions: Drug: Paclitaxel+carboplatin

INTERVENTIONS:
Drug: nab-Paclitaxel+carboplatin — Nab-P (Abraxis BioScience, LLC., Mclrose Park, IL, USA; drug license No. H20091059), 125 mg/m2, intravenous drip for 30 minutes once, on days 1 and 8, 21 days as a session for a total of 6 sessions; at the same time, carboplatin (Qilu Pharmaceutical Co., Ltd., Jinan, Shandong Province, China; drug license No. Guoji Zhunzi H20020181), AUC=2 mg•min/mL, intravenous drip for 120 minutes once, on days 1 and 8, 21 days as a session for a total of 6 sessions.
  Other Names: nab-Paclitaxel group
  Arms: nab-Paclitaxel group
Drug: Paclitaxel+carboplatin — Paclitaxel (Yangtze River Pharmaceutical Co., Ltd., Taizhou, Jiangsu Province, China; drug license No. Guoyao Zhunzi H20053001), 125 mg/m2, intravenous drip for 30 minutes once, on days 1 and 8, 21 days as a session for a total of 6 sessions; at the same time, carboplatin, AUC=2 mg•min/mL, intravenous infusion for 120 minutes once, on days 1 and 8, 21 days as a session for a total of 6 sessions.
  Other Names: Paclitaxel group
  Arms: paclitaxel group

SUMMARY:
Triple-negative breast cancer (TNBC) accounts for about 20% of clinical breast cancer. Clinical characteristics include early onset, high malignancy and heterogeneity. There is no effective drug target for TNBC, resulting in poor outcomes, high relapse rate and distant metastasis. So, further research on TNBC pathological features is particularly important.

Compared with the solvent-based paclitaxel, albumin-bound paclitaxel (nab-P) demonstrates a stronger therapeutic effect. With albumin nanoparticles as a carrier, nab-P increases the concentration of extra-tumor drugs by passing through the albumin receptor (Gp60) transmembrane pathway and the secreted protein acidic and rich in cysteine (SPARC) approach that binds to the extracellular matrix of the tumor. Numerous clinical trials have found that nab-P is superior to the solvent-based paclitaxel in the treatment of breast cancer, especially in breast cancer with poor prognosis. However, the current efficacy of nab-P in the treatment of TNBC has not been fully verified. The mechanism underlying the killing effect of nab-P on TNBC breast cancer cells remains unclear yet. This trial will compare the therapeutic effect of nab-P with solvent-based paclitaxel in TNBC patients, and seek for important scientific clues, scientific evidence, and clinical data for nab-P in the treatment of TNBC.

DETAILED DESCRIPTION:
Breast cancer has been one of the most common malignant tumors with highest morbidity and mortality that threatens women's health worldwide. Among US women, there were 250,000 new invasive breast cancers and 40,000 breast cancer deaths in 2017. In the US, 12.4% women develop breast cancer in their lifetime, and the incidence of breast cancer in women over 50 years of age has increased significantly. Although the development of molecular typing and comprehensive treatments have significantly improved the prognosis of breast cancer patients, the recurrence and metastasis of breast cancer is still the main cause of death in breast cancer patients.

TNBC accounts for about 20% of clinical breast cancer. Clinical characteristics include early onset, high malignancy and heterogeneity. There is no effective drug target for TNBC, resulting in poor outcomes, high relapse rate and distant metastasis. So, further research on TNBC pathological features is particularly important.

Paclitaxel is a natural secondary metabolite isolated and purified from the bark of Taxus chinensis. It has been clinically proven to have a good anti-tumor effect. However, polyoxyethylene castor oil/ethanol is often used as a solvent for paclitaxel in clinical practice, and this solvent-based paclitaxel is prone to causing severe allergic reactions, even aggravating myelosuppression and neurotoxicity. In addition, the solvent-based paclitaxel can also influence the efficacy of other drugs by inhibiting albumin-mediated drug delivery. nab-P is a novel paclitaxel that can compensate for the adverse effects of solvent-based paclitaxel and have good efficacy and safety. Compared with the solvent-based paclitaxel, nab-P demonstrates a stronger therapeutic effect. With albumin nanoparticles as a carrier, nab-P increases the concentration of extra-tumor drugs by passing through the albumin receptor (Gp60) transmembrane pathway and the secreted protein acidic and rich in cysteine (SPARC) approach that binds to the extracellular matrix of the tumor. Numerous clinical trials have found that nab-P is superior to the solvent-based paclitaxel in the treatment of breast cancer, especially in breast cancer with poor prognosis. However, the current efficacy of nab-P in the treatment of TNBC has not been fully verified. The mechanism underlying the killing effect of nab-P on TNBC breast cancer cells remains unclear yet.

This trial will compare the therapeutic effect of nab-P with solvent-based paclitaxel in TNBC patients, and seek for important scientific clues, scientific evidence, and clinical data for nab-P in the treatment of TNBC.

ELIGIBILITY:
Inclusion Criteria:

* breast cancer is confirmed by the mammography, and the immunohistochemical results of cancer tissues are negative for estrogen receptor, progesterone receptor and anti-human epidermal growth factor receptor 2;
* positive for axillary lymph node metastasis;
* 18-70 years of age, female;
* patients have good compliance with the planned treatment, who are volunteer to participate in the study, are willing to be treated with solvent-based paclitaxel or nab-P at random, and provide written informed consent with the premise of fully understanding the study protocol.

Exclusion Criteria:

* pregnant and lactating women;
* distant metastasis;
* patients with a history of other cancers or who have received radiotherapy on the chest;
* abnormalities in blood tests or presence of other symptoms of infection;
* allergy to paclitaxel;
* patients who have psychotropic drug abuse until now or those with a history of mental disorders;
* abnormalities in important organs such as the heart, lung, liver and kidney;
* patients who have participated in other clinical trials.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 1498 (Estimated)
Dates: Start 2021-07-19 (Estimated); Primary Completion 2025-11-30 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
Pathologic complete response (PCR) | At 5 years of treatment
  Pathologic complete remission refers to no invasive tumor cell remnants in the pathological examination of the primary mammary gland and axillary lymph nodes surgically removed. The PCR indicates the proportion of the patients with pathological complete remission to the total number of patients.

SECONDARY OUTCOMES:
Proportion of tumor stem cells in the lesion | At 9 and 18 weeks of treatment
  The CD44/CD24 expression in the breast tissues will be detected by immunohistochemistry before treatment and at 9 and 18 weeks of treatment, to determine the proportion of tumor stem cells in the lesion.
Progression-free survival (PFS) | Within 5 years of follow-up
  PFS refers to the time from random enrollment to disease progression or death for any reason indicated by imaging findings. PFS will be recorded within 5 years of follow-up.
Overall survival (OS) | Within 5 years of follow-up
  OS refers to the time from enrollment to death
Adverse events | in 5 years
  Any untoward medical occurrence in a patient and which does not necessarily have a causal relationship with this treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Caigang Liu, M.D., Ph.D., Principal Investigator — Shengjing Hospital
Locations (1):
- Shengjing Hospital of China Medical University, Shenyang, Liaoning, China